CLINICAL TRIAL: NCT01919658
Title: Effects of Femoral Versus Saphenous Nerve Blocks on Knee Extensor Strength, Pain, and Patient-Perceived Physical Function Following ACL Reconstruction
Brief Title: Effects of Femoral vs Saphenous Nerve Blocks on Function After ACL Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling, aim already examined in literature.
Sponsor: Robert A. Gallo (Other)
Responsible Party: Sponsor-Investigator, Robert A. Gallo, Assistant Professor of Orthopaedic Surgery Sports Medicine, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 42734
Record Dates: First submitted 2013-08-06; First posted 2013-08-09 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Anterior Cruciate Ligament
Keywords: nerve blocks in Anterior cruciate ligament surgery
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- proximal nerve block (Active Comparator): The anesthesiologist will administer a proximal nerve block if specified in the randomization envelope.
  Interventions: Procedure: nerve block
- distal nerve block (Active Comparator): The anesthesiologist will administer a distal nerve block if specified in the randomization envelope.
  Interventions: Procedure: nerve block

INTERVENTIONS:
Procedure: nerve block — A nerve block performed as per standard of care: femoral nerve blocks, and saphenous nerve blocks performed more distally (within 10cm superior to the adductor tubercle).

SUMMARY:
The primary objective of the study is to compare motor strength in knee extension between two groups of patients. One group receiving a proximal thigh block of the femoral nerve, and one receiving a distal thigh block of the saphenous nerve. The secondary objective is to compare the pain relief and functional outcomes in these two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Upcoming ACL reconstruction using patellar tendon autograft scheduled at Hershey Medical Center or the Hershey Outpatient Surgical Center (HOSC)

Exclusion Criteria:

1. Documented neuropathy
2. Skeletally immature
3. Previous knee surgery
4. Inability to provide informed consent
5. ACL reconstruction with other tendon repairs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
strength of knee extensors | change from baseline preoperatively at 12 months
  Extensor testing will be conducted in both legs using a hand held dynamometer.

SECONDARY OUTCOMES:
pain level and functional outcomes | change from in hospital post-operative period at 12 months
  Medical record will be reviewed for type and amount of in hospital post operative medication and levels, then assessed by PROMIS survey at follow up appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gallo, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States